CLINICAL TRIAL: NCT03516812
Title: Bipolar Androgen Therapy Plus Olaparib in Patient With Castration-Resistant Prostate Cancer
Brief Title: Testosterone and Olaparib in Treating Patients With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Michael Schweizer, Associate Professor, Division of Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9984; NCI-2018-00542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9984 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1718004 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-04-19; First posted 2018-05-04 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — olaparib; testosterone enanthate; Testosterone Propionate; testosterone 17 beta-cypionate; tetracarboxyphenylporphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (olaparib, testosterone enanthate or cypionate) (Experimental): Patients receive olaparib PO BID on days 1-28 and testosterone enanthate or cypionate IM on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Olaparib; Other: Quality-of-Life Assessment; Other: Survey Administration; Drug: Testosterone Enanthate; Drug: Testosterone Cypionate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Olaparib — Given PO
  Other Names: AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies
Drug: Testosterone Enanthate — Given IM
  Other Names: Andro LA; Androtardyl; Delatestryl; Everone; Primosteston; Testate; Testinon; Testo-Enant
Drug: Testosterone Cypionate — Given IM
  Other Names: Depo-Testosterone; TC; TCPP; Testosterone cyclopentylpropionate; Testosterone cyclopentanepropionate; Testosterone 17β-cyclopentylpropionate

SUMMARY:
This phase II trial studies how well testosterone (enanthate or cypionate) and olaparib work in treating patients with prostate cancer that has progressed despite hormonal therapy. Hormonal therapy, such as leuprolide, may lessen the amount of male sex hormones made by the body. In patients that have developed progressive cancer in spite of standard hormonal treatment (i.e. castration-resistant prostate cancer), administering testosterone may result in regression of tumors by causing DNA damage in cancer cells that have adapted to low testosterone conditions. Olaparib may stop the growth of tumor cells by blocking some of the enzymes involved in repairing DNA damage. Therefore, giving testosterone and olaparib together may work better in treating castration-resistant prostate cancer by generating DNA damage that the cancer cell is unable to repair.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the prostate-specific antigen (PSA)50 response rate (i.e., percent of patients with a PSA decline of at least 50% below baseline) following 12-weeks of treatment with bipolar androgen therapy (BAT) plus olaparib in men with asymptomatic metastatic castration-resistant prostate cancer (mCRPC) who have progressed on abiraterone and/or enzalutamide.

SECONDARY OBJECTIVES:

I. Determine the percent of mCRPC patients achieving a radiographic response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria following treatment with BAT plus olaparib.

II. Determine the radiographic progression free survival (PFS) in mCRPC patients treated with BAT plus olaparib using RECIST 1.1 criteria for soft tissue metastases and Prostate Cancer Working Group 3 (PCWG3) criteria for bone metastases.

III. Determine the PSA PFS rate according to PCWG3 criteria in mCRPC patients treated with BAT plus olaparib.

IV. Determine the PFS (i.e. whichever occurs first: clinical, radiographic or PSA progression) in mCRPC patients treated with BAT plus olaparib.

V. Determine the overall survival in mCRPC patients treated with BAT plus olaparib.

VI. Track changes in quality of life (QoL) as determined using the Functional Assessment of Cancer Therapy -Prostate (FACT-P) and International Index of Erectile Function (IIEF) surveys.

VII. Assess the incidence and severity of adverse events according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

EXPLORATORY OBJECTIVES:

I. Evaluate for differences in response and PFS in patients with/without mutations in genes involved in homologous recombination.

II. Determine intratumoral androgen levels using liquid chromatography-mass spectrometry (LC/MS).

III. Assess for evidence of double stranded deoxyribonucleic acid (dsDNA) breaks using gamma-H2AX immunostaining on circulating tumor cells (CTCs) and metastatic tissue.

IV. Assess androgen receptor (AR) and AR splice variant (AR-V) transcript expression levels using quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) on CTCs.

V. Assess androgen receptor (AR) and AR splice variant (AR-V) protein expression levels using immunostaining on circulating tumor cells (CTCs) and metastatic tissue.

VI. Sequence tumor DNA (cell-free circulating tumor DNA [ctDNA] and/or metastatic tissue).

VII. Conduct transcript profiling studies on CTCs (multiplexed qRT-PCR) and metastatic tissue (ribonucleic acid sequencing [RNA-seq]).

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28 and testosterone enanthate or cypionate intramuscularly (IM) on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients are followed up at 30 days and every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to provide informed consent prior to any study specific procedures
* Documented histologically confirmed adenocarcinoma of the prostate
* Patient must have evidence of castration resistant prostate cancer as evidenced by PSA progression (per Prostate Cancer Working Group 3 [PCWG3] criteria) and a castrate serum testosterone level (i.e., ≤ 50 mg/dL)
* PSA must be at least 1 ng/ml and rising on two successive measurements at least two weeks apart
* Patients must have progressed on abiraterone and/or enzalutamide; there must be at least a 3-week washout period after stopping the most recent approved therapy for mCRPC (i.e., abiraterone, enzalutamide, Ra-223, sipuleucel-t); if applicable, patients should be weaned off steroids at least 1 week prior to starting treatment
* No prior chemotherapy for the treatment of mCRPC; patients may have received docetaxel for the treatment of hormone-sensitive prostate cancer
* Prior treatment with non-chemotherapy investigational agents is permitted; there must be at least a 3-week washout period after stopping any investigational cancer agent
* Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (within 28 days prior to administration of study treatment)
* Platelet count ≥ 100 x 10^9/L (within 28 days prior to administration of study treatment)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5 x ULN (within 28 days prior to administration of study treatment)
* Patients must have creatinine clearance estimated using the Cockcroft-Gault equation or based on a 24 hour urine test of ≥ 51 mL/min (within 28 days prior to administration of study treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have a life expectancy ≥ 16 weeks
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by computed tomography (CT), positron-emission tomography (PET), magnetic resonance imaging (MRI) and/or bone scan and is suitable for repeated assessment
* Must have archival tissue available, be willing to undergo metastatic biopsy or have a sufficient plasma circulating tumor DNA (ctDNA) concentration in order to perform next-generation DNA sequencing
* The study will require that 50% of enrolled subjects have homozygous deletions, deleterious mutations, or both in one or more of the DNA damage response (DDR) genes; the other 50% of patients must have an intact DDR pathway

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment in this study
* Participation in another clinical study with an investigational product during the last 3 weeks
* Any previous treatment with poly-adenosine diphosphate ribose polymerase (PARP) inhibitor, including olaparib
* Other malignancy unless curatively treated with no evidence of disease for ≥ 5 years except: adequately treated non-melanoma skin cancer
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, Fridericia's corrected QT interval [QTcF] prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil); the required washout period prior to starting olaparib is 2 weeks
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil); the required washout period prior to starting olaparib is 3 weeks for enzalutamide, 5 weeks for phenobarbital and 3 weeks for other agents
* Persistent toxicities (> Common Terminology Criteria for Adverse Event [CTCAE] grade 2) caused by previous cancer therapy, excluding alopecia
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Patients with symptomatic uncontrolled brain metastases; a scan to confirm the absence of brain metastases is not required; the patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment; patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection; examples include, but are not limited to, uncontrolled ventricular arrhythmia, history of prior myocardial infarction, uncontrolled major seizure disorder, uncontrolled hypertension (blood pressure [BP] ≥ 160/100), history of prior stroke, uncontrolled diabetes (glycosylated hemoglobin [hgb A1C] > 7), unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product
* Patients with a known hypersensitivity to the testosterone cypionate or any of the excipients of the product
* Patients with known active hepatitis (i.e., hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable)
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule
* Evidence of disease that, in the opinion of the investigator, would put the patient at risk from testosterone therapy (e.g. femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction)
* Patients with pain attributable to their prostate cancer
* Tumor causing urinary outlet obstruction that requires catheterization for voiding; patients that require catheterization to void secondary to benign strictures or other non-cancer causes will be permitted to enroll
* Prior history of deep venous thrombosis or pulmonary embolism within 5 years prior to enrollment in the study and not currently on systemic anticoagulation
* Patients with NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) prior to enrollment in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Started | 36
Completed | 30
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 70.1 [51.8 to 87.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 9
PSA [Median (Full Range); unit: ng/ml] | 25.6 [2.2 to 1409.7]
Prior abiraterone treatment [Count of Participants; unit: Participants] | 25
Prior enzalutamide treatment [Count of Participants; unit: Participants] | 18
Prior docetaxel treatment [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With a Prostate-specific Antigen (PSA) Decline of at Least 50% Below Baseline PSA50 Response Rate
Description: PSA response will be defined as a decline in PSA ≥ 50% compared to baseline in patients who received at least 12 weeks of treatment. Will be calculated as the percentage with 95% confidence interval (CI) of the total number of subjects that achieved a PSA response.
Time Frame: Median time to PSA50 response was 22 weeks.
Population: Includes patient that received at least 12 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 30
Participants | 14

2. Secondary Outcome: Incidence of Adverse Events (AEs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03
Description: Number of patients experiencing an adverse event
Time Frame: Up to 30 days after last dose, 19 month median
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 36
Participants | 33

3. Secondary Outcome: Radiographic Response Rate
Description: Per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines, a radiographic response (as determined on CT or MRI) will be defined as: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 13
Participants | 8

4. Secondary Outcome: PSA Progression Free Survival (PFS)
Description: Median time to PSA progression free survival in months with 95% CI
Time Frame: Up to 2 years following the last dose of study drug, median of 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 36
months | 7 [4 to 11]

5. Secondary Outcome: Overall Survival (OS)
Description: Median overall survival in months with 95% CI will be calculated.
Time Frame: Up to 2 years following the last dose of study drug, median 29 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 36
months | 26 [22 to 99999]

6. Secondary Outcome: Radiographic PFS
Description: Median radiographic progression free survival in months with 95% CI.
Time Frame: Up to 2 years following the last dose of study drug, median 19 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 36
months | 13 [7 to 17]

7. Secondary Outcome: Average Change in Quality of Life (QOL) Assessed by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) Survey
Description: Average change in total Functional Assessment of Cancer Therapy-Prostate (FACT-P) quality of life (QOL) score after 4 cycles of treatment. FACT-P is a validated survey designed to assess the QOL in patients with prostate cancer. The FACT-P contains 39 items that use a 0-4 rating scale. The highest possible score is 156 (lowest possible score = 0). The total score is an indication of overall quality of life, where the higher scores indicate better quality of life.Score is reported as units on a scale.
Time Frame: From baseline and up to 5 years after initiating therapy, median 19 months
Population: Number of patients who completed FACT-P QOL survey after 4 cycles of treatment.
Measure: Mean (95% Confidence Interval); unit: Mean differences in score
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 22
Mean differences in score | 1.36 [-4.89 to 7.33]

8. Secondary Outcome: Average Change in Quality of Life (QOL) Assessed by the International Index of Erectile Function (IIEF) Survey
Description: Participants were assessed using the International Index of Erectile Function (IIEF) which is a validated multidimensional scale for erectile function and ejaculatory function in men. The questionnaire consists of 3 questions with a scale for each from 0-5 (highest overall score 15, lowest score 0). The higher the score, the better the outcome and vice versa. Score is reported as units on a scale.
Time Frame: Up to 5 years after initiating therapy, median 19 months
Population: Number of patients who completed IIEF QOL survey after 4 cycles of treatment.
Measure: Mean (95% Confidence Interval); unit: Mean differences in score
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
Number analyzed (Participants) | 22
Mean differences in score | 2.56 [-0.93 to 6.04]

ADVERSE EVENTS:
Time Frame: Serious and other AEs assessed for up to 2 years and within 30 days of stopping study drugs, median 19 months
Arm/Group | Treatment (olaparib, testosterone enanthate or cypionate)
All-Cause Mortality (participants affected / at risk) | 2/36
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 33/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (olaparib, testosterone enanthate or cypionate) (N=36)
Subdural hematoma (Nervous system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Rib fracture (Musculoskeletal and connective tissue disorders) | 1
Stroke (Nervous system disorders) | 1
Cord compression (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (olaparib, testosterone enanthate or cypionate) (N=36)
Fatigue (General disorders) | 21
Nausea (Gastrointestinal disorders) | 18
Pain (General disorders) | 13
Constipation (Gastrointestinal disorders) | 8
Anemia (Blood and lymphatic system disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Dysgeusia (Nervous system disorders) | 5
Creatinine increase (Renal and urinary disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness or Lightheadedness (Nervous system disorders) | 3
Nocturia (Renal and urinary disorders) | 3
Weight loss (Metabolism and nutrition disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Edema (Blood and lymphatic system disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Insomnia (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Thromboembolic event (Vascular disorders) | 2
Urinary retention (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03516812/Prot_SAP_000.pdf